CLINICAL TRIAL: NCT00245414
Title: Post-marketing Clinical Trial of Pegasys® 180μg for Subcutaneous Injection in Patients With Chronic Hepatitis C. General Clinical Study in Interferon (IFN)-Treated and IFN-untreated Chronic Hepatitis C Patients, Except for Those Infected With High Viral Load of Genotype 1b
Brief Title: Trial of Pegasys® in Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical, Chugai Pharmaceutical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18501
Record Dates: First submitted 2005-10-27; First posted 2005-10-28 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2010-11

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Interferon (IFN)-Treated
  Interventions: Drug: Pegasys®
- 2 (Experimental): Interferon (IFN)-Untreated and Quantitative serum HCV-RNA is positive at week 1
  Interventions: Drug: Pegasys®
- 3 (Experimental): Interferon (IFN)-Untreated and Quantitative serum HCV-RNA is negative at week 1
  Interventions: Drug: Pegasys®
- 4 (Experimental): Interferon (IFN)-Untreated and Quantitative serum HCV-RNA is negative at week 1
  Interventions: Drug: Pegasys®

INTERVENTIONS:
Drug: Pegasys® — 180μg for s.c./week for 48 weeks
  Arms: 1; 2; 3
Drug: Pegasys® — 180μg for s.c./week for 24 weeks
  Arms: 4

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of Pegasys® 180μg for subcutaneous (s.c.) injection in interferon (IFN)-treated or IFN-untreated chronic hepatitis C patients except for those infected with genotype 1b of hepatitis C virus (HCV) and a high viral load (≥ 100 KIU/mL).

In addition, this study will explore the efficacy and safety of Pegasys® 180μg for s.c. injection given at 2 different periods between 24 and 48 weeks in IFN-untreated chronic hepatitis C patients.

ELIGIBILITY:
Inclusion Criteria:

* Quantitative serum HCV-RNA is positive except for high viral load of genotype 1b (≥ 100 KIU/mL)
* Observation of serum ALT elevation above upper limit of normal
* Chronic hepatitis is evaluated as the negative result (< 0) calculated by the method of "formula for discrimination between chronic hepatitis and liver cirrhosis."

Exclusion Criteria:

* Observation of white blood cells ≦ 3000/mm3; neutrophils ≦ 1500/mm3; platelets ≦ 90,000/mm3; or hemoglobin ≦ 10 g/dL.
* Observation of the following situations and disease: severe renal disease, hepatitis B co-infection, de-compensated liver disease, liver cirrhosis, hepatocellular carcinoma, poorly controlled psychiatric disease, seizure disorders, immunologically mediated disease, severe cardiac disease, poorly uncontrolled hypertension, poorly controlled diabetes, chronic pulmonary disease, retinopathy, malignant tumor, and organ transplant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2005-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Sustained viral response as undetectable level of HCV-RNA | week 24 from the end of treatment

SECONDARY OUTCOMES:
Biochemical response as normal level of ALT | week 24 from the end of treatment
Viral response as undetectable level of HCV-RNA | at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ken Kashima, Study Director — Chugai Pharmaceutical
Locations (6):
- Japan (6):
  - Kyusyu Region, Fukuoka
  - Chugoku Region, Okayama
  - Kinki Region, Osaka
  - Hokkaido Region, Sapporo
  - Kanto Region, Tokyo
  - Tokai Region, Yamanashi